CLINICAL TRIAL: NCT07211399
Title: The Role of Intraoperative Opioids in the Transition From Acute to Chronic Opioid Use and Chronic Pain
Brief Title: Transition From Acute to Chronic Opioid Use and Chronic Pain
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25050099
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a prospective RCT aiming to examine the effectiveness of OFA on the reduction of postoperative acute and chronic pain and opioid use among 700 adult TKA patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-free anesthesia (OFA) Group (Experimental): Subjects enrolled in this arm will receive IV-acetaminophen, IV-lidocaine, dexmedetomidine, and ketamine prior to intubation.
  Interventions: Drug: Opioid-free anesthesia
- Opioid-based anesthesia (OBA) Group (Active Comparator): Subjects enrolled in this arm will receive IV-acetaminophen, IV-lidocaine, and fentanyl prior to intubation.
  Interventions: Drug: Opioid-based anesthesia

INTERVENTIONS:
Drug: Opioid-free anesthesia — Each patient will be pre-oxygenated receive IV-acetaminophen (1 g), and IV-lidocaine (60 - 100 mg). and dexmedetomidine (12-20 mcg IV) and ketamine (25-50 mcg) prior to intubation. Induction of anesthesia will be achieved with IV-propofol (1 - 2 mg/kg; 150 - 200 mg). Patient air ways will be secured with an intratracheal tube or LMA. Anesthesia will be maintained by either propofol (100 - 150 mcg/kg/hour; TIVA), or sevoflurane (0.5-1 MAC). During surgery, dexmedetomidine and ketamine will be administered as needed. Anesthesia will be maintained by either propofol (100 - 150 mcg/kg/hour; TIVA), or sevoflurane (0.5-1 MAC).
  Other Names: Dexmedetomidine & Ketamine Group
  Arms: Opioid-free anesthesia (OFA) Group
Drug: Opioid-based anesthesia — Each patient will be pre-oxygenated receive IV-acetaminophen (1 g), and IV-lidocaine (60 - 100 mg). and fentanyl 50-100 mcg IV prior to intubation. Induction of anesthesia will be achieved with IV-propofol (1 - 2 mg/kg; 150 - 200 mg). Patient air ways will be secured with an intratracheal tube or LMA. Anesthesia will be maintained by either propofol (100 - 150 mcg/kg/hour; TIVA), or sevoflurane (0.5-1 MAC). During surgery, each patient in the opioid group will receive IV-fentanyl (50 - 100 mcg) as needed.
  Other Names: Fentanyl Group
  Arms: Opioid-based anesthesia (OBA) Group

SUMMARY:
In the current opioid crisis, the use of opioids as the main pain management method is recognized as a consistent risk factor for chronic opioid use and the development of Opioid Use Disorder (OUD), as well as related complications like overdose fatalities among surgical patients. The most recent data suggests that 3.1%-10.5% of surgical patients are at risk of developing OUD. On average, there are over 40 million major surgeries that require post-op pain management, taking place in the United States each year. This puts over 1 million American surgical patients at risk for opioid dependency and misuse.

This is a prospective randomized controlled intervention study that will examine the physical and emotional outcomes of surgical patients who receive intraoperative Opioid-Free Anesthesia (OFA) supplemented with Non-Opioid Analgesia (NOAs), and how this relates to surgical patients who receive intraoperative Opioid-Based Anesthesia (OBA).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* scheduled for an elective, unilateral Total Knee Arthroplasty (TKA)
* anticipated to stay in PACU after surgery
* receiving general anesthesia (i.e. fentanyl, etc.)
* receiving spinal regional anesthesia

Exclusion Criteria:

* <18 years of age
* sent to the ICU at any point during their hospital stay
* scheduled for a bilateral TKA
* received intraoperative opioids other than fentanyl
* received patient-controlled analgesia in PACU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
PACU Opioid Medication Administered | Postoperative Day 5
  Medications will be extracted from the electronic medical records. Opioid-based medications will be reported as mean(SD).
PACU Non-Opioid Medication Administered | Postoperative Day 5
  Medications will be extracted from the electronic medical records.Non-opioid-based medications will be reported as mean(SD).
PACU NRS Pain Score at Rest | Postoperative Day 5
  Numerical Rating Scale (NRS) Pain Scores will be self reported on a scale of 0-10, 0 being no pain at all, 10 being worst pain imaginable. Pain scores at rest will be averaged and reported as mean(SD).
PACU NRS Pain Score with Movement | Postoperative Day 5
  Numerical Rating Scale (NRS) Pain Scores will be self reported on a scale of 0-10, 0 being no pain at all, 10 being worst pain imaginable. Pain scores with movement will be averaged and reported as mean(SD).

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Chelly, MD, PhD, MBA, Principal Investigator — University of Pittsburgh, UPMC
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified information collected throughout the study will be included in a study database. No patient identifiers will be included in the database and there will be a confidential (access limited to investigators only) code or link between the database and other information about the participant. De-identified data may be shared with additional internal or external data warehouses/investigators and the NIH.
  Data may be shared with authorized representatives of the study sponsor and federal regulatory agencies for purposes of monitoring the conduct of this study.
  If data is to be shared with other external organizations in the future, the IRB will be modified accordingly, and an appropriate Date Use Agreement will be secured.